CLINICAL TRIAL: NCT00270309
Title: Self-management for Men With Uncomplicated Lower Urinary Tract Symptoms. A Randomised Controlled Trial Against Standard Therapy
Brief Title: Self-management for Men With Uncomplicated Lower Urinary Tract Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Royal College of Surgeons of England (Other)
Collaborators: University College, London (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 64582
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2005-12

CONDITIONS: Uncomplicated Lower Urinary Tract Symptoms
Keywords: lower urinary tract symptoms, self-management
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Self-Management

INTERVENTIONS:
Behavioral: Self-management

SUMMARY:
Objective To test the hypothesis that a nurse-led self-management programme is effective for men with uncomplicated lower urinary tract symptoms. This will be achieved by comparing symptom seveirty and the amount of drug therapy used to manage these symptoms in men who attend a self-management programme, compared to those who do not.

Study design This study will use the format of a randomised controlled trial. 200 new patients with uncomplicated LUTS will be randomised to either attend or not attend (standard therapy) a self-management programme. The programme provides education, reassurance, prostate cancer risk, advice on lifestyle modifications (e.g. fluids - type and amount), concurrent medication re-scheduling and behavioural changes (double-voiding, strategies for dribbling, and bladder re-training). These strategies are learnt through group discussion, problem solving and goal setting.

All men start the study with a period of watchful waiting (monitoring symptoms only) and are followed up for a total of 1 year. At each assessment (baseline, 3, 6, and 12 months) symptom severity and the use of drug therapy to control symptoms will be compared between the two groups. The only difference between them is that one group has attended a self-management programme and the other has not.

Potential application of results Self-management focuses on patient involvement in health care by involving them in the day-to-day control of their symptoms. If effective, self-management may provide a long-term method of managing LUTS without using drug therapy, thereby offering considerable health gain and financial savings.

The NHS Modernisation Agency wishes to develop the role of the nurse specialist to manage some patients independently of doctors. Nurse-led LUTS assessment clinics are now well established, perhaps nurses managing these patients with self-management interventions may become part of standard therapy.

DETAILED DESCRIPTION:
1. OBJECTIVES

   To assess the effectiveness of self-management interventions in men with uncomplicated LUTS.
2. STUDY DESIGN

   2.1 This is a randomised controlled trial comparing self-management with standard therapy. These interventions are proposed to optimise watchful waiting, providing an alternative to drugs and surgery for symptom control.

   Participants

   2.2. Participating urological units include the Middlesex Hospital NHS Trust and the Whittington Hospital NHS Trust.

   2.3. 200 new patients with uncomplicated LUTS (I-PSS score 0-35) will be randomised to either attend a self-management programme or not attend a self-management programme (standard therapy - control group). There will be approximately 100 men in each group. Standard therapy, as described previously, involves watchful waiting, drugs or surgery, the therapeutic choice depending on weighting severity and bother, with risks and benefits.

   2.4. All new patients over the age of 40 years with a diagnosis of lower urinary tract symptoms secondary to benign prostatic hyperplasia or age related bladder dysfunction are eligible for inclusion.

   2.5. The following exclusion criteria applies:
   * age under 40 yrs
   * lower urinary tract symptoms due to any urological malignancy or whilst investigating any urological malignancy e.g. prostate cancer
   * previous prostatic surgery within the last 10 years or pelvic radiotherapy
   * complications of urinary obstruction (acute or chronic urinary retention - post micturition volumes over 300ml, bladder stones, renal failure, recurrent urinary tract infection or haematuria)
   * uncontrolled diabetes, dementia and end stage cardiac or respiratory failure
   * inability to speak or understand the English language
   * severe symptoms where drug therapy or surgical management is indicated or requested by the patient
   * any man who is or has been in the previous 3 months on medical therapy for lower urinary tract symptoms, including alpha-blockers, 5-alpha reductase inhibitors (finasteride) or anti-cholinergics. The use of alpha-blockers for the control of hypertension is permitted, since these men have symptoms and still are eligible for medical treatment (finasteride, anti-cholinergics) and surgery.

   2.6. Each patient will be fully informed regarding the study process and possible uses of subsequent data collected. An information sheet on headed paper will be available and a consent form signed by both researcher and patient. The patients who participate in this study will not participate in any other study conducted by our group in the future.

   2.7. All GP's will be informed by letter of their patient's participation and progress in this study. A copy of this standard letter will be left in the patients' notes on recruitment.

   2.8. Once recruited men will be randomised into 2 groups. Computer generated randomisation will be carried out by a third party. Randomisation takes place at week zero of each mans 12 months overall participation in the study. Patients will be recruited by the study coordinator. On recruitment an enrolment form is completed, and a copy left in the patient notes along with their consent form.

   2.9. Group 1 will receive self-management and Group 2 will receive standard therapy.

   2.10. All men start the study with a period of watchful waiting until their first assessment at 2 months. During this time men assigned to self-management will attend their 3 sessions, the control group will not.

   2.11. Men in Groups 1 & 2 will be followed up as per protocol at 2, 6, and 12 months after randomisation i.e. short, medium, and long term.

   Intervention

   2.12. Men randomised into Group 1 (self-management) will in addition to standard follow up, be invited to attend 3 small group (4-6 men) sessions and receive a single telephone call (as their self-management programme).

   2.13. The four key areas within the self-management programme are:
   * Education
   * Reassurance
   * Lifestyle modifications
   * Behavioural changes

   2.14. The sessions will be facilitated by local nurse practitioners).

   2.15. The sessions are standardised and run from a Facilitators Manual developed and piloted at The Royal College of Surgeons and The Centre for Behavioural and Social Sciences in Medicine, UCL.

   2.16. Each session lasts approximately 2 hours and is a mixture of group learning through brainstorming and discussion, teaching, and goal setting. All sessions are supported with a self-management booklet given in session 1.

   2.17. Session 1 (first week):
   * Introduction and programme review
   * Introduction to the concept of self-management
   * Education/reassurance - prostate and bladder health, prostate cancer, future symptoms
   * Managing fluid intake
   * Caffeine abstinence
   * Alcohol advice

   2.18. Session 2 (second week):
   * Adjusting medications which affect LUTS e.g. diuretics (if relevant)
   * Constipation advice
   * Strategies for dribbling
   * Double-voiding
   * Bladder re-training

   2.19. Third week telephone call - trouble shooting problems and answering queries

   2.20. Session 3 (six weeks):
   * Booster session
   * Designed for men to share reasons why some things work and others do not
   * Used to discuss reasons why for example they have found it difficult to abstain from caffeine or other goals set

   2.21. Each man in Group 1 will be able to contact the Clinical Nurse Specialist at other times aside from the sessions in the case of confusion or query, by telephone, e-mail or letter.

   Intervention components

   2.22. Education - Men with LUTS should understand:
   * LUTS are real symptoms worthy of medical care
   * Not all LUTS require treatment with drugs and/or surgery (give details of expected future symptomology)
   * That patients have an important role to play in the management of their symptoms
   * Each patient has the ability to follow a self-management programme which can have a beneficial effect on their symptoms - self-efficacy
   * The range of treatments available for men with LUTS including why some treatments are used and not others i.e. the appropriateness of treatment

   2.23. Reassurance - Men with LUTS should understand:
   * The symptom severity of many men with LUTS does not change over time (85% stable at 1 year and 65% at 5 years [17,18])
   * Some men may see spontaneous symptom improvement
   * The annual risk of acute urinary retention is 2% [19]
   * LUTS are often affected by a man's current state of mind, high levels of arousal or worry can have a detrimental effect
   * Their symptoms are not due to detectable prostate cancer
   * That their risk of prostate cancer is that of an age related man with no symptoms i.e. that of the general male population of the same age [20]

   2.24. Lifestyle modifications include fluid, caffeine and alcohol advice.

   Fluid advice • Introduce the concept of a healthy fluid balance
   * Explain the significance of concentrated urine and the potential detrimental (irritative) effects
   * There are good fluid habits all men can use regularly with minimal effort
   * There are specific changes that some men may have to make based on their previously completed charts e.g. excessive intake of water at night
   * Excessive or inadequate fluid intake should always be avoided
   * A total daily intake of 1500-2000 mls is advised (minor adjustments made for climate and activity)
   * Fluid should be spaced evenly throughout the day rather than in large single amounts
   * Fluid restriction for symptom control at times of greatest inconvenience e.g. long car journeys or when out in public places, is appropriate, but the overall daily intake should not be restricted significantly (for control of irritative symptoms)
   * If nocturia is bothersome, fluid restriction 2 hours before retiring to bed can be effective

   Caffeine Advice

   • Explain that caffeine has a detrimental effect on symptoms in men with LUTS especially irritative symptoms
   * Explain that caffeine can be found in tea, coffee, chocolate, energy drinks and over the counter flu remedies
   * Explain that by completely avoiding caffeine, symptom improvement may be found
   * If caffeine use is excessive then it should not be stopped overnight but over 2-3 days to avoid headaches and stomach cramps etc
   * Caffeine avoidance can be achieved by substituting for drinks that are de-caffeinated or non-caffeinated e.g. de-caffeinated coffee or a soft drink
   * Nocturia can be exacerbated by evening caffeine use, to prevent this caffeine should be avoided for 5 hours prior to retiring

   Alcohol advice

   • Explain that alcohol has a detrimental effect on symptoms in men with LUTS especially irritative symptoms

   • Explain that by completely avoiding alcohol, symptom improvement may be found, but that we understand this may not be possible and avoiding alcohol or restriction of alcohol at times of greatest inconvenience may be more appropriate
   * Explain there are quality of life issues with alcohol abstinence and this information is a guide only
   * In men with nocturia evening alcohol use should be avoided
   * Explain when we consume alcohol we often consume large quantities of extra fluid and symptom reduction may be achieved by substituting large volume alcoholic drinks for small volume alcoholic drinks e.g. a pint to a short

   Timing of concurrent medication • Adjust the time medication (with an effect on urinary symptoms) is taken to improve LUTS at times of most inconvenience e.g. meetings, long car journeys and when out in public places

   • Substitute an anti-hypertensive diuretic (with the aid of the patient's GP) to a suitable alternative with less urinary effects in a man with LUTS

   Behavioural changes • Men with obvious 'bad habits' will be advised e.g. the going 'just in case' type of man

   • Men with LUTS will be advised to double void

   • Men with post micturition dribble should be advised on urethral milking

   • Men with LUTS who have 'irritative' symptoms will be offered a formal bladder re-training programme.

   • Advice will be given to men with LUTS regarding avoiding constipation

   2.25. Men randomised to the self-management arm of the study will also be offered a booster or refresher session at six-months, or just after their six month assessment.

   Outcomes

   2.26. The primary outcome is treatment failure. In this study treatment failure is defined as:

   • The use of drug therapy for symptom control (as determined by a consultation between clinician and patient)
   * Surgical intervention (as determined by a consultation between clinician and patient)
   * Symptom deterioration of 3 points[22] or more measured with the I-PSS
   * Acute urinary retention
   * Death

   2.27. Secondary outcomes include a 3 day frequency / volume chart, infection, and health-seeking behaviour (unscheduled clinic, A&E or GP visits). Secondary outcomes also include Quality of life / bother assessment using the BPH Impact Index,[24] (appendix 5.), Short Form-36 - SF-36 (appendix 7.) and the Illness Perception Questionnaire - IPQ (appendix 8.).

   The clinicians will be blinded to which group the patients have been assigned to, and the patients will be asked not to divulge which group they are in. It is not possible to blind the patients to the group to which group they are assigned to. Any instances of unblinding will be declared.

   Follow up assessment

   2.28. Men within the study group will see only the consultant or the specialist registrar (i.e. continuity throughout the study) doctors will be briefed to the study design but blinded as to which group each man has been assigned to.

   2.29. If a man has deteriorated significantly then drug therapy (alpha-blockers, finasteride or anti-cholinergics) will be offered; standard urological practice. As these men will only see one of 2 different doctors, moving from conservative to drug therapy will be consistent.

   2.30. The outcome of the consultation between clinician and patient will be recorded by the clinician on a standard form (appendix 9.) and given to the patient, a copy will be left in the notes.

   2.31. At this visit the patient will be given the following to complete: I-PSS, BPH Impact Index, SF-36, Illness perception questionnaire and a 3-day frequency / volume chart, and will be asked to send to the data manager along with the outcome form completed by the consultant in a pre-paid envelope.

   2.32. The data manager is blinded to which group the patient is in and will be responsible for collecting, loading, and chasing missing data. The data manager will telephone each patient within 48 hours of their out-patient follow up to complete the assessment and encourage completion of the study documents.

   2.33. A follow up rate of more than 80% will be achieved.

3. STATISTICAL ANALYSIS

3.1. The two groups will be directly compared with respect to all outcome measurements over each man's 12 month study period.

3.2. Analysis will be on an intention to treat basis, i.e. - men will always be analysed in the group to which they were assigned.

3.3. Statistical analysis will be performed with STATA Version 7. An unpaired t-test will be used to analyse continuous variables e.g. I-PSS, and chi-squared or exact tests will be used for categorical data. Logarithmic transformation will be used to normalise continuous variables.

3.4. Sample size - A minimum of 84 men are required in each group to have a 90% chance of detecting a 3 point difference in mean I-PSS score (SD=6) at the 5% level of significance using the unpaired t-test. We have chosen a 3-point reduction in I-PSS as it corresponds to a detectable clinical difference in symptoms by patients.

4. DATA COLLECTION

4.1. Each man is part of the study programme for 12 months. After this time each man is discharged from the study programme. If they still require the services of the urology out-patients for further appointments, investigations or treatment, this will be arranged.

4.2. If self-management is seen to be effective then it will be offered to men in Group 2 who received only standard treatment.

4.3. The information is anonymised with each patient being given a unique identification number.

4.4. Data will be stored securely on The Royal College of Surgeons network in accordance with the Data Protection Act 1988. Access to this data will be limited to the data manager and the study coordinator

ELIGIBILITY:
Inclusion Criteria:

* new patients with uncomplicated LUTS (I-PSS score 0-35)
* aged 40 years and over
* referred for the first time by their family doctor (general practitioner) to one of a participating urological outpatient departments

Exclusion Criteria:

* lower urinary tract symptoms due to any urological malignancy
* previous prostatic surgery within the last 10 years or pelvic radiotherapy
* complications of urinary obstruction (acute or chronic urinary retention - post micturition volumes over 300ml, bladder stones, renal failure, recurrent urinary tract infection or haematuria)
* uncontrolled diabetes, dementia and end stage cardiac or respiratory failure
* inability to speak or understand the English language
* severe symptoms where drug therapy or surgical management is indicated or requested by the patient
* medical therapy for lower urinary tract symptoms in the previous 3 months, including alpha-blockers, 5-alpha reductase inhibitors (finasteride) or anti-cholinergics.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168
Dates: Start 2004-01; Primary Completion 2004-04 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
treatment failure (use of drug therapy for symptom control, surgical intervention, symptom deterioration of 3 points or more measured with the I-PSS, acute urinary retention, or death)

SECONDARY OUTCOMES:
quality of life / bother assessment (BPH Impact Index)
Short Form-36
Illness Perception Questionnaire - IPQ
health-seeking behaviour (unscheduled clinic, A&E or GP visits)
infection
3 day frequency / volume chart

CONTACTS AND LOCATIONS:
Overall Officials: Christian Brown, Principal Investigator — Clinical Effectiveness Unit, The Royal College of Surgeons of England; Mark Emberton, Study Chair — Clinical Effectiveness Unit, The Royal College of Surgeons of England; Jan HP Van der Meulen, PhD, Study Director — Clinical Effectiveness Unit, The Royal College of Surgeons of England

REFERENCES:
- [Background] Brown CT, van der Meulen J, Mundy AR, O'Flynn E, Emberton M. Defining the components of a self-management programme for men with uncomplicated lower urinary tract symptoms: a consensus approach. Eur Urol. 2004 Aug;46(2):254-62; discussion 263. doi: 10.1016/j.eururo.2004.02.008. PMID 15245822
- [Background] Brown CT, Van Der Meulen J, Mundy AR, Emberton M. Lifestyle and behavioural interventions for men on watchful waiting with uncomplicated lower urinary tract symptoms: a national multidisciplinary survey. BJU Int. 2003 Jul;92(1):53-7. doi: 10.1046/j.1464-410x.2003.04268.x. PMID 12823383
- [Background] Newman S, Steed L, Mulligan K. Self-management interventions for chronic illness. Lancet. 2004 Oct 23-29;364(9444):1523-37. doi: 10.1016/S0140-6736(04)17277-2. PMID 15500899
- [Derived] Brown CT, Yap T, Cromwell DA, Rixon L, Steed L, Mulligan K, Mundy A, Newman SP, van der Meulen J, Emberton M. Self management for men with lower urinary tract symptoms: randomised controlled trial. BMJ. 2007 Jan 6;334(7583):25. doi: 10.1136/bmj.39010.551319.AE. Epub 2006 Nov 21. PMID 17118949
- See also: Project list of the Clinical Effectiveness Unit, The Royal College of Surgeons of England — http://www.rcseng.ac.uk/surgical_research_units/ceu/projects/index.html
- See also: Centre for Behavioural and Social Sciences in Medicine, University College London, UK — http://www.ucl.ac.uk/medicine/